CLINICAL TRIAL: NCT05561465
Title: Evaluation of Pterygomaxillary Disjunction With Interpositional Y-shape Plate as an Innovative Minimally Invasive Technique in Patients With Temporomandibular Joint Internal Derangement (Clinical Trial)
Brief Title: Pterygomaxillary Disjunction With Interpositional Y-shape Plate in Patients With Temporomandibular Joint Derangement
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hams Hamed Abdelrahman (Other)
Responsible Party: Sponsor-Investigator, Hams Hamed Abdelrahman, Assistant lecturer of DPH and Clinical statistician, Alexandria University
Organization: Alexandria University (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TMD_2021
Record Dates: First submitted 2022-09-27; First posted 2022-09-30 (Actual); Last update posted 2022-09-30 (Actual); Status verified 2022-09

CONDITIONS: Temporomandibular Disorder
MeSH Terms: conditions — Temporomandibular Joint Disorders

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Pterygomaxillary disjunction (Experimental)
  Interventions: Procedure: Pterygomaxillary disjunction with interposition Y-shape plate

INTERVENTIONS:
Procedure: Pterygomaxillary disjunction with interposition Y-shape plate — All patients will be treated under general anesthesia. The pterygoid plate will be fractured, pried up, and pushed backward. A Y-shape plate will be fixed to the lateral maxillary surface with its vertical limb and the other two limbs are turned to fit into the retro maxillary space preventing the reattachment of the fractured pterygoid plate

SUMMARY:
Temporomandibular joint internal derangement (TMJ ID) is the most frequent type of temporomandibular disorder (TMDs)which is managed by different therapeutic modalities. it begins with conservative methods like medical treatment, physiotherapy, thermotherapy, and bites appliance therapy. Surgical intervention is a controversial issue in cases not responding to conservative methods. A novel minimally invasive surgical technique which is extracapsular trans oral (Pterygomaxillary disjunction) has been advocated as a minimally invasive extracapsular technique that preserves TMJ integrity.

ELIGIBILITY:
Inclusion Criteria:

* Patients without relevant disease
* Patients refractory to conservative treatment > 6 months.
* Patients are diagnosed, with unilateral/bilateral anterior disc displacement without reduction, clinically and by MRI recently.
* No previous TMJ surgery.
* No previous maxillofacial trauma.

Exclusion Criteria:

* Patients with systemic joint disease (rheumatoid, osteoarthritis, gouts).
* Medically compromised patients contraindicating operation.
* Patients to whom general anesthesia is contraindicated.
* Patient with neuromuscular disorders.
* Patients with any gross pathology of the ear.
* Patient with psychoneurotic disorders.

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 12 (Actual)
Dates: Start 2021-11-01 (Actual); Primary Completion 2022-06-30 (Actual); Study Completion 2022-06-30 (Actual)

PRIMARY OUTCOMES:
Change in wound healing | 1st week and 2nd week
  The sutured wounds will be examined after one and two weeks for signs and symptoms of infection including swelling, redness, hotness, pus discharge, and pain in addition to observation for any manifestations of wound healing disturbance, as wound dehiscence and hardware exposure.
Change in TMJ clinical dysfunction | 1st week, 2nd week, 1 month, and 3 months
  Helkimo's dysfunction index is used, including the interincisal opening of the mandible, deviation during the opening, dysfunction of TMJ, pain in the TMJ and preauricular region, and also masticatory muscles were palpated for pain during the follow-up periods.
disc position | at 3 months
  MRI assessment by proton-density (PD), Evaluation by MRI will be done after 3 months to assure disc position.

CONTACTS AND LOCATIONS:
Locations (1):
- Outpatient Clinic of Oral and Maxillofacial Surgery Department, Faculty of Dentistry, Alexandria University, Alexandria, Egypt